CLINICAL TRIAL: NCT06344624
Title: Comparing Brief Cognitive-behavioral Group Therapy and Laughter Yoga on Depression and Psychological Resilience in Nursing Students With Mental Symptoms: A Randomized Controlled Trial
Brief Title: The Effect of Cognitive and Laughter Therapy on Psychological Symptoms in Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Emine ÖNCÜ, Assoc.Prof, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Mersin_U
Record Dates: First submitted 2024-03-25; First posted 2024-04-03 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Mental Health Issue
Keywords: Brief cognitive-behavioral group therapy; laughter yoga; mental symptoms; nursing students

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial with a pretest-posttest design
Who Masked: Participant, Outcomes Assessor
Masking Description: Using the block randomization technique, the sampled students will be split into two groups: the CBT group and the laughter group. Six will be the block size. Excel will be used to create blocks (allocation concealment) and random numbers will be generated by an assistant researcher who does not attend therapy sessions. The purpose of the program is to support mental health and evaluate its effectiveness; students will not be informed about which group they are in (participant blinding).
  Research data will be coded as A and B and entered into the computer database by someone other than the researchers conducting the therapy sessions, and statistical analysis will be performed using this coding (statistician blinding).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Behavioral Therapy Group (Active Comparator): In the first sessions, less time was allotted to the introductory phase because it was anticipated that students would face similar issues in terms of age, gender, and academic standing, and that their depressive symptoms would be milder than those of clinical patient groups. Additionally, more intensive short-term cognitive behavioral therapy (b-CBT) was preferred. Six sessions, two per week for three weeks, lasting sixty minutes each, were planned, with four groups of eight to twelve students based on course schedules. A researcher with a doctorate in mental health nursing and certification in CBT will oversee CBT. The program aims to enhance students' mindful awareness. Key CBT techniques will include breath-body awareness, coping methods for emotional and physical depression symptoms (breathing and attention exercises), recognizing thought-emotion-behavior interactions, cognitive restructuring, and future planning.
  Interventions: Behavioral: CBT group
- Laughter Yoga Therapy Group (Active Comparator): There will be a certified researcher leading the laughter yoga sessions. Laughter yoga will ideally allow participants to sit comfortably in front of each other's eyes. Six sessions, two per week for three weeks, lasting sixty minutes each, were planned, with four groups of eight to twelve students based on course schedules. Laughter yoga consists of four parts: deep breathing exercises, warm-up exercises, playful activities, and laughter exercises.
  Interventions: Behavioral: Laughter group

INTERVENTIONS:
Behavioral: CBT group — Brief cognitive behavioral therapy
  Arms: Cognitive Behavioral Therapy Group
Behavioral: Laughter group — Laughter yoga therapy
  Arms: Laughter Yoga Therapy Group

SUMMARY:
The presence of high mental symptoms among nursing students in Turkey highlights the need to develop various support strategies in nursing education to preserve and ensure the continuity of the nursing workforce. This study aims to compare the effects of brief cognitive-behavioral group psychotherapy and laughter yoga on mental symptoms in nursing students with mental symptoms.

DETAILED DESCRIPTION:
A randomized controlled trial with a pretest-posttest design is planned to be conducted among 114 nursing students with mental symptoms between April and June 2024. The block randomization method will be used to assign students to the Cognitive Behavioral Therapy (CBT) Group and the Laughter Group. Brief cognitive behavioral therapy (b-CBT) will be applied to one group, and laughter yoga will be applied to the other group twice a week for 3 weeks, with sessions lasting 60 minutes each. Data will be collected through the Brief Symptom Inventory, Psychological Resilience Scale, and Automatic Thoughts Scale. Measurements will be done at baseline, right after the sixth session ends, and four weeks later.

During the b-CBT process, techniques such as breath-body awareness and self-identification, coping techniques for emotional and physical symptoms of depression, recognizing the interaction between thoughts, emotions, and behaviors, cognitive restructuring to replace dysfunctional thoughts and internal dialogues with functional ones, and future planning will be employed. Laughter yoga will consist of four parts: deep breathing exercises, warm-up exercises, playful activities, and laughter exercises.

The results obtained from the research will provide an opportunity to identify methods that may be effective in helping nurses acquire the necessary skills to improve their mental health.

ELIGIBILITY:
Inclusion Criteria:

Currently enrolled in the nursing faculty between April 10, 2024, and June 2, 2024.

* Scored within the top 20% on the Brief Symptom Inventory for mental symptom scores.
* Voluntarily agree to participate in the study and have signed the Informed Consent Form.
* Understand and comprehend Turkish language

Exclusion Criteria:

* Having received cognitive behavioral therapy previously.
* Undergoing psychological or psychiatric treatment.
* Underwent surgical procedures in the last three months.
* Having chronic illnesses requiring regular medication use.
* Having glaucoma or hernia conditions.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 114 (Actual)
Dates: Start 2024-04-10 (Actual); Primary Completion 2024-06-02 (Actual); Study Completion 2024-06-12 (Actual)

PRIMARY OUTCOMES:
The change in mental symptoms will be assessed using the Brief Symptom Inventory. | Changing from at baseline (pretest- T0) and right after the end of the 6th season (post test- T1) and and 4 weeks later the end of the 6th season (T2).
  The scale consists of 53 Likert-type items. Items are scored on a scale of 0 to 4, corresponding to "not at all" and "very much," respectively. The higher the total score obtained from the scale, the more the individual's mental symptoms increase. It comprises nine subscales, three global indices, and additional items. The subscales are somatization, obsessive-compulsive disorder, interpersonal sensitivity, depression, anxiety disorder, hostility, phobic anxiety, paranoid ideation, and psychoticism, while additional items relate to eating disorders, sleep disturbances, thoughts of death and suicide, and feelings of guilt.

SECONDARY OUTCOMES:
Psychological resilience will be assessed using the Psychological Resilience Scale. | Changing from at baseline (pretest- T0) and right after the end of the 6th season (post test- T1) and 4 weeks later the end of the 6th season (T2).
  The Psychological Resilience Scale (PRS) consists of six items that respondents self-report on a 5-point Likert scale. Higher scores correspond to higher psychological resilience levels. The scores for items 2, 4, and 6 are reversed. The response options on the Likert scale range from "not at all suitable" (1), "not suitable" (2), "somewhat suitable" (3), "suitable" (4), and "completely suitable" (5). With an internal consistency score of.83, the scale has a high Cronbach's alpha coefficient.
Negative self-evaluations and thought patterns will be assessed using the Automatic Thoughts Scale. | Changing from at baseline (pretest- T0) and right after the end of the 6th season (post test- T1) and 4 weeks later the end of the 6th season (T2).
  This scale is designed to measure common thought patterns and negative self-evaluations often seen in depression. The scale is in Likert format and consists of 30 items. For each item, response options range from "never" (1), "rarely" (2), "occasionally" (3), "frequently" (4), and "always" (5). A higher score denotes a higher frequency of automatic thoughts linked to depression. The total score ranges from 30 to 150. The Cronbach's α coefficient for the scale is 0.95.

CONTACTS AND LOCATIONS:
Overall Officials: EMİNE ÖNCÜ, Principal Investigator — Mersin University
Locations (1):
- Turkey, Mersin University, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data may be shared upon request from the principal investigator, subject to the appropriateness of the request, while ensuring adherence to the rules of confidentiality regarding individual data.
Supporting Information: Study Protocol
Time Frame: October through December of 2024
Access Criteria: Individual participant data may be shared upon request from the principal investigator, subject to the appropriateness of the request, while ensuring adherence to the rules of confidentiality regarding individual data.